CLINICAL TRIAL: NCT07201285
Title: Ultrasound-Guided Edge of Laminar Block Versus Erector Spinae Plane Block for Postoperative Analgesia in Patients Undergoing Video-Assisted Thoracoscopic Surgery: A Randomized Clinical Trial
Brief Title: Edge of Laminar Block Versus Erector Spinae Plane Block for Postoperative Analgesia in Video-Assisted Thoracoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1336/8/25
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Edge of Laminar Block; Erector Spinae Plane Block; Postoperative Analgesia; Video-Assisted Thoracoscopic Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELB group (Experimental): Patients will receive edge of laminar block using 20ml of bupivacaine 0.25%.
  Interventions: Other: Edge of laminar block
- ESPB group (Experimental): Patients will receive an erector spinae plane block using 20ml of bupivacaine 0.25%.
  Interventions: Other: Erector spinae plane block

INTERVENTIONS:
Other: Edge of laminar block — Patients will receive edge of laminar block using 20ml of bupivacaine 0.25%.
  Arms: ELB group
Other: Erector spinae plane block — Patients will receive an erector spinae plane block using 20ml of bupivacaine 0.25%.
  Arms: ESPB group

SUMMARY:
This study aims to compare the ultrasound-guided edge of laminar block (ELB) and erector spinae plane block (ESPB) for postoperative analgesia in patients undergoing video-assisted thoracic surgery (VATS).

DETAILED DESCRIPTION:
Postoperative pain after thoracic surgery, which is attributed to muscle incisions, rib retractions, and intercostal nerve damage, may be severe enough to cause pulmonary complications, such as atelectasis, pneumonia, and increased oxygen consumption.

The erector spinae plane block (ESPB) is used for managing post-thoracotomy pain and has numerous advantages that make it an attractive alternative technique. The ESPB injects a local anaesthetic around the erector spinae muscle at approximately the level of the T5. It may be able to block the dorsal and ventral rami of the thoracic spinal nerves.

A novel technique of retrolaminar block (RLB) called the edge of laminar block (ELB) to provide sensory analgesia during rib fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Undergoing video-assisted thoracic surgery (VATS) under general anesthesia.

Exclusion Criteria:

* History of allergies to local anesthetics.
* Opioid dependency.
* Bleeding or coagulation disorders.
* Psychiatric and neurological disorder.
* Local infection at the site of injection.
* Severe heart, lung, liver, and renal dysfunction.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS)> 3 to be repeated after 30 min if pain persists until the NRS < 4.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to first dose of morphine administrated).
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 0.5 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded preoperatively, before performing of block, and every 15 min till the end of surgery.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively, before performing of block, and every 15 min till the end of surgery.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at post-anesthesia care unit (PACU), 2, 4, 6, 8, 12, 18, and 24 h postoperatively.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, pruritus, urinary retention, itching, constipation, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.